CLINICAL TRIAL: NCT05392075
Title: COVID-19 Breakthrough Infection in Fully Vaccinated People and in People Who Received a Booster Dose
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 014.IMD.2022.D
Record Dates: First submitted 2022-05-24; First posted 2022-05-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 diagnosis: The study will enroll all subjects who received care at Methodist Dallas Medical Center between August 1, 2021 and February 28, 2022, and were diagnosed with COVID-19. COVID-19 diagnosis for the purpose of this study is either a positive COVID-19 antigen or a positive COVID-19 PCR test.
  Interventions: Biological: Pfizer COVID-19 mRNA vaccine; Biological: Moderna COVID-19 mRNA vaccine

INTERVENTIONS:
Biological: Pfizer COVID-19 mRNA vaccine — vaccinated people who received the Pfizer COVID-19 mRNA vaccine
Biological: Moderna COVID-19 mRNA vaccine — vaccinated people who received the Moderna COVID-19 mRNA vaccine vaccine

SUMMARY:
A novel coronavirus, SARS-CoV-2 (formerly known as the 2019 novel coronavirus [2019-nCoV]) was identified as the agent that caused an outbreak of pneumonia (termed COVID-19) in Wuhan, China in December 2019. The virus quickly spread to other countries and on March 11, 2020, the World Health Organization (WHO) declared COVID-19 a pandemic. By March 2021, many nations and organizations embarked on finding a cure or vaccine for this devastating viral infection. The Pfizer COVID-19 mRNA vaccine was the first to obtain emergency use authorization (EUA) from the Food & Drug Administration (FDA) on December 11, 2020, followed by the Moderna COVID-19 mRNA vaccine on December 18, 2020, and the Janssen COVID-19 viral vector vaccine on February 27, 2021. The mRNA vaccines and the viral vector vaccine are designed based on the spike protein of SARS-COV-2. These vaccines had been administered to millions of Americans prior to July 2021.

DETAILED DESCRIPTION:
A novel coronavirus, SARS-CoV-2 (formerly known as the 2019 novel coronavirus [2019-nCoV]) was identified as the agent that caused an outbreak of pneumonia (termed COVID-19) in Wuhan, China in December 2019. The virus quickly spread to other countries and on March 11, 2020, the World Health Organization (WHO) declared COVID-19 a pandemic. By March 2021, many nations and organizations embarked on finding a cure or vaccine for this devastating viral infection. The Pfizer COVID-19 mRNA vaccine was the first to obtain emergency use authorization (EUA) from the Food & Drug Administration (FDA) on December 11, 2020, followed by the Moderna COVID-19 mRNA vaccine on December 18, 2020, and the Janssen COVID-19 viral vector vaccine on February 27, 2021. The mRNA vaccines and the viral vector vaccine are designed based on the spike protein of SARS-COV-2. These vaccines had been administered to millions of Americans prior to July 2021.

Similar to other infections that are preventable with vaccination, COVID-19 vaccination is not a SARS-CoV-2 infection panacea. However, in fully vaccinated people the risk of SARS-CoV-2 infection, hospitalization, severe illness, and death from COVID-19 is relatively less. Viruses may escape the host immune defense through mutations that create new variants of the primary virus. Some variants emerge and disappear while others persist and may have properties that may be different from the primary virus. By late 2020, a new variant, the delta variant, was identified in Maharashtra, India. This variant is highly transmissible and causes infections even in fully vaccinated people, it is less sensitive to neutralizing antibodies from recovered subjects and less sensitive to vaccine-induced antibodies, and there is evidence that it causes more severe infections. While the world was trying to contain and control the spread of the delta variant, the WHO reported a new variant of COVID-19, omicron. It was detected in late November 2021 in specimens collected in Botswana and South Africa. New variants of SARS-CoV-2 are expected to continue to emerge and the world continues to seek means of controlling the pandemic.

COVID-19 vaccination data from the Centers for Disease Control and Prevention (CDC) showed that the population ratios who have received a full series of COVID-19 vaccination from Pfizer, Moderna, or Janssen as of February 2, 2022 is 17.46/11.25/1. Furthermore, more of those who received the Janssen COVID-19 viral vector vaccine have preferred and received an mRNA vaccine booster. Unfortunately, the CDC data lacks the booster dose data for Texas residents.

The FDA in collaboration with the CDC makes decision on when a booster is recommended. This decision is based on many factors including the level of antibodies and memory cells post-COVID-19 vaccination and infection. There is much evidence that decreasing the COVID-19 spike antibodies titer and memory cells may increase the likelihood of a breakthrough COVID-19 infection. Unfortunately, there isn't a prior report or study comparing the incidence of COVID-19 infection among people fully vaccinated with any of the approved COVID-19 vaccines. This study seeks to find a relationship between the last dose of a COVID-19 vaccine in a fully vaccinated person and a COVID-19 breakthrough infection. The study will also find a correlation between the duration from a booster dose to the diagnosis of a breakthrough COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, ≥18 years of age
* Be willing and able to provide informed consent if needed; in cases where an abbreviated telephone informed consent needs to be obtained, the patient must understand and speak English.
* Has received at least two doses of an mRNA vaccine or one dose of the Janssen COVID-19 vaccine
* Had a positive COVID-19 antigen or PCR test at least 14 days after the last COVID-19 vaccine.
* Patients who had a diagnosis of COVID-19 at a Methodist Facility within the last 30 days preceding their admission must have the result in their electronic medical record.

Exclusion Criteria:

* Does not satisfy all of the inclusion criteria.
* The patient had a COVID-19 infection diagnosed at a non-Methodist facility within the last 30 days.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All subjects who received care at Methodist Dallas Medical Center between August 1, 2021 and February 28, 2022, and were diagnosed with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Incidence rate of COVID-19 breakthrough infections in fully vaccinated | up to 6 months
  The number of COVID-19 breakthrough infections in fully vaccinated participants
incidence rate of COVID-19 breakthrough infections in fully vaccinated subjects who received a COVID-19 booster vaccine different form their initial two doses (for a mRNA vaccine) or the single-dose Janssen COVID-19 vaccine. | up to 6 months
  Comparison of the number of COVID-19 breakthrough infections in fully vaccinated subject who received a COVID-19 booster

CONTACTS AND LOCATIONS:
Overall Officials: Valentine Ebuh, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No